CLINICAL TRIAL: NCT05240378
Title: Preoperative Screening for COVID-19 and Strict COVID Cancer Protocol Helps to Reduce Postoperative Infection, Mortality and Morbidity in Cancer Patients Undergoing Surgery. A Comparative Study
Brief Title: Mortality of Cancer Surgery During SARS CoV2 Pandemic
Status: Completed | Type: Observational
Sponsor: Banaras Hindu University (Other)
Responsible Party: Principal Investigator, Manoj Pandey, Professor, Banaras Hindu University
Other Study IDs: Dean/2021/EC/3004
Record Dates: First submitted 2022-02-12; First posted 2022-02-15 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: SARS CoV 2 Infection; Cancer
MeSH Terms: conditions — COVID-19; Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre covid: Cases operated one year prior to the date of declaration of corona pandemic in India
  Interventions: Other: Surgery
- post covid: cases operated from the date of declaration of corona pandemic to one year after
  Interventions: Other: Surgery

INTERVENTIONS:
Other: Surgery — Surgery for cancer as per the stage of the disease and protocol

SUMMARY:
The impact of cancer surgery during covid epidemic is not clear. The published reports show contradictory findings that extend from no change in mortality to increased mortality, further no data on exposure and outcome of health care worker is available. This study is designed to address the above questions

DETAILED DESCRIPTION:
This is a retrospective study from the prospectively collected data that is extracted from the electronic database of Department of Surgical Oncology, IMS, BHU The data is inform of two cohorts one extending from April 2019-April 2020 and other from May 2020 to May 2021 i.e. pre covid and during covid pandemic

ELIGIBILITY:
Inclusion Criteria:

* All patients operated during the study period

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All cases of cancer operated between April 2019 to May 2021
Sampling Method: Non-Probability Sample
Enrollment: 1576 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
30 day mortality | 30 days
  post operative deaths within one year
number of participants developing major or minor complications | 30 days
  Surgical complications classified as per Clavien Dindo classification

SECONDARY OUTCOMES:
number of health care worker with SARS CoV2 infection | 1 year
  Covid infection in health care workers

CONTACTS AND LOCATIONS:
Overall Officials: Manoj Pandey, MS, PhD, Principal Investigator — Banaras Hindu University
Locations (1):
- Banaras Hindu University, Varanasi, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared on reasonable request as per Indian law